CLINICAL TRIAL: NCT03666832
Title: Multi-center, Open-label, Phase 1b Clinical Trial to Evaluate the Safety, Tolerability, and Exploratory Efficacy of TEW-7197 in Combination With FOLFOX in Patients With Metastatic Pancreatic Ductal Adenocarcinoma Who Have Failed First-Line Gemcitabine and Nab-Paclitaxel
Acronym: MP-PDAC-01
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Joon Oh Park (Other)
Responsible Party: Sponsor-Investigator, Joon Oh Park, Samsung Medical Center, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-10-150
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm1 (Experimental): TEW-7197 100mg will be administered orally once a day 5days and rest 2days. Study treatment will be continued until objective disease progression.
  Interventions: Drug: TEW-7197

INTERVENTIONS:
Drug: TEW-7197 — TEW-7197 1cycle 14days
  -intake 5days, rest 2days
  Other Names: TEW-7197, FOLFOX

SUMMARY:
* Inclusion

  1. Subjects who are males or females ≥ 19 years of age
  2. Subjects who have the following history of first-line gemcitabine and nab-paclitaxel among patients with cytologically or histologically proven metastatic pancreatic ductal adenocarcinoma
  3. Subjects who can give written informed consent for participation in this trial after receiving explanations of this trial
  4. Subjects who have the following laboratory test values:

     * bilirubin ≤ 1.5 x ULN (upper limit of normal)
     * aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 x ULN
     * serum creatinine ≤ 1.5 x ULNor estimated creatinine clearance ≥ 40 mL/min (Cockcroft-Gault)
     * partial thromboplastin time (aPTT) ≤ 1.5 x ULN
     * absolute neutrophil count (ANC) ≥ 1,500 cells/µL
     * platelet count ≥ 100,000/µL
     * hemoglobin ≥ 9.0 g/dL
  5. Subjects who have at least a 12-week life expectancy at the Investigator's discretion
  6. Subjects who have Eastern Cooperative Oncology Group (ECOG)Performance Status 0-1
* Exclusion

  1. Subjects who were treated with surgery, radiotherapy, chemotherapy or investigational therapy within 2 weeks (note: placement of biliary stent is allowed)
  2. Subjects who have uncontrolled CNS metastases (patients who require steroids should be on a stable or decreasing dose for at least 2 weeks)
  3. Subjects who have any contraindications for 5-FU, leucovorin, or oxaliplatin
  4. Subjects who have moderate or severe cardiovascular disease

     * Subjects who have myocardial infarction, unstable angina pectoris, New York Heart Association (NYHA) Class III/IV congestive heart failure, or uncontrolled hypertension within 6 months before screening
     * Subjects who have major abnormalities at the Investigator's discretion based on electrocardiogram (ECG)and Doppler ECHO results at screening or within 14 days before screening
     * Subjects who have increase in brain natriuretic peptide(BNP) or increase in troponin (over 99th percentile upper reference limit) at Screening (based on the normal range of relevant study center)
     * Subjects who have risk factors for ascending aortic aneurysm such as genetic disorder and trauma and risk factors for aortic stenosis
     * Subjects who have a history of heart or aorta surgery
  5. Subjects who have clinically significant gastrointestinal bleeding within 4 weeks before screening
  6. Subjects who have a known history or suspected hypersensitivity to any excipients of the investigational product or combination drug(s)
  7. Subjects who have received prior treatment targeting the signaling pathway of TGF-β
  8. Subjects who have a disease or condition that affects the mechanism of the investigational product, or are currently using or planning to use:

     * Drugs that are exclusively or primarily eliminated by cytochrome P-450 isozyme (CYP) including CYP1A2, CYP2B6, or CYP3A4
     * Drugs that are exclusively or primarily eliminated by UDP glucuronyltransferase (UGT) 1A1 (UGT1A1)
     * Drugs that are substrates for the drug transporter multidrug resistance protein 1 (MDR1) have a narrow therapeutic window or are strong inhibitors of drug transporter MDR1
     * Drugs that are strong inhibitors or inducers of CYP2D6 or CYP3A4
  9. Subjects who are unable to swallow tablets
  10. Subjects who have a history of or are suspected of drug abuse
  11. Female subjects of child-bearing potential who have a positive result on a pregnancy test at screening or are unable to agree to use an effective barrier method of birth control to avoid pregnancy during the study period (e.g., sterilization, intrauterine contraceptive device, combination of oral contraception and barrier contraception, combination of other hormone delivery systems and barrier contraception, contraceptive cream, combination of cream, jelly, or form and diaphragm or condom)
  12. Subjects, in the opinion of the Investigator, who are unsuitable to participate in the study
  13. Subjects who were treated with other investigational products within 28 days before screening or within a period shorter than 5-timesthe half-life of the investigational product

ELIGIBILITY:
Inclusion Criteria:

* 1) Subjects who are males or females ≥ 19 years of age 2) Subjects who have the following history of first-line gemcitabine and nab-paclitaxel among patients with cytologically or histologically proven metastatic pancreatic ductal adenocarcinoma 3) Subjects who can give written informed consent for participation in this trial after receiving explanations of this trial 4) Subjects who have the following laboratory test values:
* bilirubin ≤ 1.5 x ULN (upper limit of normal)
* aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 x ULN
* serum creatinine ≤ 1.5 x ULNor estimated creatinine clearance ≥ 40 mL/min (Cockcroft-Gault)
* partial thromboplastin time (aPTT) ≤ 1.5 x ULN
* absolute neutrophil count (ANC) ≥ 1,500 cells/µL
* platelet count ≥ 100,000/µL
* hemoglobin ≥ 9.0 g/dL 5) Subjects who have at least a 12-week life expectancy at the Investigator's discretion 6) Subjects who have Eastern Cooperative Oncology Group (ECOG)Performance Status 0-1

Exclusion Criteria:

* 1) Subjects who were treated with surgery, radiotherapy, chemotherapy or investigational therapy within 2 weeks (note: placement of biliary stent is allowed) 2) Subjects who have uncontrolled CNS metastases (patients who require steroids should be on a stable or decreasing dose for at least 2 weeks) 3) Subjects who have any contraindications for 5-FU, leucovorin, or oxaliplatin 4) Subjects who have moderate or severe cardiovascular disease
* Subjects who have myocardial infarction, unstable angina pectoris, New York Heart Association (NYHA) Class III/IV congestive heart failure, or uncontrolled hypertension within 6 months before screening
* Subjects who have major abnormalities at the Investigator's discretion based on electrocardiogram (ECG)and Doppler ECHO results at screening or within 14 days before screening
* Subjects who have increase in brain natriuretic peptide(BNP) or increase in troponin (over 99th percentile upper reference limit) at Screening (based on the normal range of relevant study center)
* Subjects who have risk factors for ascending aortic aneurysm such as genetic disorder and trauma and risk factors for aortic stenosis
* Subjects who have a history of heart or aorta surgery 5) Subjects who have clinically significant gastrointestinal bleeding within 4 weeks before screening 6) Subjects who have a known history or suspected hypersensitivity to any excipients of the investigational product or combination drug(s) 7) Subjects who have received prior treatment targeting the signaling pathway of TGF-β 8) Subjects who have a disease or condition that affects the mechanism of the investigational product, or are currently using or planning to use:
* Drugs that are exclusively or primarily eliminated by cytochrome P-450 isozyme (CYP) including CYP1A2, CYP2B6, or CYP3A4
* Drugs that are exclusively or primarily eliminated by UDP glucuronyltransferase (UGT) 1A1 (UGT1A1)
* Drugs that are substrates for the drug transporter multidrug resistance protein 1 (MDR1) have a narrow therapeutic window or are strong inhibitors of drug transporter MDR1
* Drugs that are strong inhibitors or inducers of CYP2D6 or CYP3A4 9) Subjects who are unable to swallow tablets 10) Subjects who have a history of or are suspected of drug abuse 11) Female subjects of child-bearing potential who have a positive result on a pregnancy test at screening or are unable to agree to use an effective barrier method of birth control to avoid pregnancy during the study period (e.g., sterilization, intrauterine contraceptive device, combination of oral contraception and barrier contraception, combination of other hormone delivery systems and barrier contraception, contraceptive cream, combination of cream, jelly, or form and diaphragm or condom) 12) Subjects, in the opinion of the Investigator, who are unsuitable to participate in the study 13) Subjects who were treated with other investigational products within 28 days before screening or within a period shorter than 5-timesthe half-life of the investigational product

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-06-17 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
pregression free survival | up to 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea